CLINICAL TRIAL: NCT01274975
Title: Safety of Autologous Adipose Derived Mesenchymal Stem Cells in Patients With Spinal Cord Injury
Brief Title: Autologous Adipose Derived MSCs Transplantation in Patient With Spinal Cord Injury.
Acronym: MSC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Astrostem
Record Dates: First submitted 2011-01-06; First posted 2011-01-12 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Other: Autologous Adipose Derived Mesenchymal Stem Cells — Intravenous infusion of Autologous Adipose Derived Mesenchymal Stem Cells. Dose : 4 x 10e8 cells
  Other Names: Astrostem®

SUMMARY:
This study is designed to assess the safety of intravenous autologous adipose derived mesenchymal stem cells transplant in spinal cord injury patients.

DETAILED DESCRIPTION:
Adipose derived mesenchymal stem cells (AdMSCs) represent an attractive and ethical cell source for stem cell therapy.

With the recent demonstration of MSC homing properties, intravenous aplications of MSCs to cell-damaged diseases have increased.

In a human clinical trial, eight male patients who had suffered a spinal cord injury were intravenously administered autologous hAdMSCs (4×10e8 cells) one time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and sign the consent form for this study.
* Age :19-60, males
* Clinical diagnosis of spinal cord injury(American Spinal Injury Association[ASIA] Impairment Scale[AIS] grade A or B or C)
* Duration of injury : > 2 months

Exclusion Criteria:

* Subjects who must put on a respirator
* Subjects who had malignant tumor within 5 years
* Subjects with a infectious disease include HIV and hepatitis
* Subjects who injured brain or spinal cord before spinal cord injury
* Subjects who has high body temperature more than 38℃ or acute disorder
* Subjects with anemia or thrombocytopenia
* Subjects with angina pectoris, myocardial infarction, cardiomyopathy, occlusive disease, chronic renal failure, glomerular disease and chronic obstructive pulmonary disease
* Subjects with congenital or acquired immunodeficiency disorders
* Subjects with muscular dystrophy or articular rigidity
* Patients with clouded consciousness or speech disorder
* treat with cytotoxic medications(immunosuppressive drug, corticosteroid and cytotoxic drug) during clinical trials
* participating another clinical trials within 3 months
* other serious disease or disorder that could seriously affect ability to participate in the study

Ages: 19 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
safety evaluation | 12weeks
  Safety evaluate through physical examination, vital sign and laboratory test after "RNL-Astrostem" injected

CONTACTS AND LOCATIONS:
Overall Officials: SangHan Kim, MD, Principal Investigator — Anyang Sam Hospital

REFERENCES:
- [Result] Ra JC, Shin IS, Kim SH, Kang SK, Kang BC, Lee HY, Kim YJ, Jo JY, Yoon EJ, Choi HJ, Kwon E. Safety of intravenous infusion of human adipose tissue-derived mesenchymal stem cells in animals and humans. Stem Cells Dev. 2011 Aug;20(8):1297-308. doi: 10.1089/scd.2010.0466. Epub 2011 Mar 17. PMID 21303266